CLINICAL TRIAL: NCT01810926
Title: A Phase II Multicentre, Randomized, Controlled Open-label Study on the Use of Anti-thymocyte Globulin and Rituximab for Immunomodulation of Graft-versus-host Disease in Allogeneic Matched Transplants for Non Malignancies
Brief Title: T&B Depletion Non Malignant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Franco Locatelli (Other)
Collaborators: University of Milano Bicocca (Other); medac GmbH (Industry); Fresenius AG (Industry)
Responsible Party: Sponsor-Investigator, Franco Locatelli, Director Department of Pediatric Hematology and Oncology, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPBG_361.11; 2011-004730-34 (EudraCT Number)
Record Dates: First submitted 2012-01-16; First posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Graft Versus Host Disease
Keywords: indication for HSCT; matched related donor; MRD; Matched Unrelated Donor; MUD
MeSH Terms: conditions — Graft vs Host Disease | interventions — Rituximab; treosulfan; fludarabine; fludarabine phosphate; Thiotepa; Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MRD-Regimen&Polyclonal antibody (Experimental): Patients MRD will be randomized to receive Treosulfan iv at a dose of 14 g/m² within 120 minutes on day -7, - 6, -5 + Fludarabine iv at a dose of 30 mg/ m² within 30 minutes on day -7, -6, -5,-4,-3 after treosulfan + Thiotepa iv at a dose of 8 mg/kg on day - 3 divided into 2 infusions at 12 hrs intervals + Cyclosporine A iv at a dose of 3 mg/kg/day starting from day -1 and a dose adjustment will be done to obtain plasma levels of 150-250 ng/mL + Methotrexate iv at a dose of 15 mg/m2 on day +1, at a dose of 10 mg/m2 on day + 3 and + 6 & ATG-Fresenius S® iv at a dose of 5 mg/kg within 8 hours on day -4,-3,-2
  Interventions: Biological: polyclonal antibody; Drug: Treosulfan; Drug: Fludarabine; Drug: Thiotepa; Drug: Cyclosporine A; Drug: Methotrexate
- MRD-Regimen (Sham Comparator): Patients receiving stem cell transplantation from a matched related donors (MRD) will be randomized to receive only Treosulfan iv at a dose of 14 g/m² within 120 minutes on day -7, - 6, -5 (total dose of 42 g/m²) + Fludarabine iv at a dose of 30 mg/ m² within 30 minutes on day -7, -6, -5,-4,-3 (total dose of 150 mg/m²) after treosulfan + Thiotepa iv at a dose of 8 mg/kg on day - 3 divided into 2 infusions at 12 hrs intervals (total dose of 8 mg/kg)+ Cyclosporine A iv at a starting dose of 3 mg/kg/day starting from day -1 and a dose adjustment will be done to obtain plasma levels of 150-250 ng/mL (In the absence of GvHD CSA will be tapered after day + 180 and stopped at 9-12 months) + Methotrexate iv at a dose of 15 mg/m2 on day +1, at a dose of 10 mg/m2 on day + 3 and + 6
  Interventions: Drug: Treosulfan; Drug: Fludarabine; Drug: Thiotepa; Drug: Cyclosporine A; Drug: Methotrexate
- MUD-Regimen & Rituximab (Experimental): Patients MUD will be randomized to receive Treosulfan iv at a dose of 14 g/m² within 120 minutes on day -7, - 6, -5 + Fludarabine iv at a dose of 30 mg/ m² within 30 minutes on day -7, -6, -5,-4,-3 after treosulfan + Thiotepa iv at a dose of 8 mg/kg on day - 3 divided into 2 infusions at 12 hrs intervals + Cyclosporine A iv at a dose of 3 mg/kg/day starting from day -1 and a dose adjustment will be done to obtain plasma levels of 150-250 ng/mL + Methotrexate iv at a dose of 15 mg/m2 on day +1, at a dose of 10 mg/m2 on day + 3 and + 6 and at a dose of 10 mg/m2 on day +11 + ATG-Fresenius S ® iv at a dose of 5 mg/kg within 8 hours on day -4,-3,-2 & Rituximab in a single infusion of 200 mg/m2 on day -1
  Interventions: Biological: polyclonal antibody; Drug: Rituximab; Drug: Treosulfan; Drug: Fludarabine; Drug: Thiotepa; Drug: Cyclosporine A; Drug: Methotrexate
- MUD-Regimen (Sham Comparator): Patients MUD will be randomized to receive only Treosulfan iv at a dose of 14 g/m² within 120 minutes on day -7, - 6, -5 + Fludarabine iv at a dose of 30 mg/ m² within 30 minutes on day -7, -6, -5,-4,-3 after treosulfan + Thiotepa iv at a dose of 8 mg/kg on day - 3 divided into 2 infusions at 12 hrs intervals + Cyclosporine A iv at a dose of 3 mg/kg/day starting from day -1 and a dose adjustment will be done to obtain plasma levels of 150-250 ng/mL + Methotrexate iv at a dose of 15 mg/m2 on day +1, at a dose of 10 mg/m2 on day + 3 and + 6 and at a dose of 10 mg/m2 on day +11 + ATG-Fresenius S ® iv at a dose of 5 mg/kg within 8 hours on day -4,-3,-2
  Interventions: Biological: polyclonal antibody; Drug: Treosulfan; Drug: Fludarabine; Drug: Thiotepa; Drug: Cyclosporine A; Drug: Methotrexate

INTERVENTIONS:
Biological: polyclonal antibody — iv at a dose of 5 mg/kg within 8 hours on day -4,-3,-2 (total dose 15 mg/kg)
  Other Names: ATG S Fresenius
  Arms: MRD-Regimen&Polyclonal antibody; MUD-Regimen; MUD-Regimen & Rituximab
Drug: Rituximab — single infusion of200 mg/m2 on day -1
  Other Names: Mabthera
  Arms: MUD-Regimen & Rituximab
Drug: Treosulfan — iv at a dose of 14 g/m² within 120 minutes on day -7, - 6, -5 (total dose of 42 g/m²)
  Other Names: Medac
Drug: Fludarabine — iv at a dose of 30 mg/ m² within 30 minutes on day -7, -6, -5,-4,-3 after treosulfan
  Other Names: Fludara
Drug: Thiotepa — iv at a dose of 8 mg/kg on day - 3 divided into 2 infusions at 12 hrs intervals
  Other Names: Tepadina
Drug: Cyclosporine A — iv at a dose of 3 mg/kg/day starting from day -1 and a dose adjustment will be done to obtain plasma levels of 150-250 ng/mL
  Other Names: Neoral
Drug: Methotrexate — iv at a dose of 15 mg/m2 on day +1, at a dose of 10 mg/m2 on day + 3 and + 6
  Arms: MRD-Regimen; MRD-Regimen&Polyclonal antibody
Drug: Methotrexate — iv at a dose of 15 mg/m2 on day +1, at a dose of 10 mg/m2 on day + 3 and + 6 and at a dose of 10 mg/m2 on day +11
  Arms: MUD-Regimen; MUD-Regimen & Rituximab

SUMMARY:
• The primary aim of the present trial is to assess in a randomized fashion the benefit on standard graft-versus-host disease (GVHD) prophylaxis of the addition of ATG-Fresenius S ® in transplants from matched related donors (MRD) and of anti-CD20 rituximab in transplants from matched unrelated donors (MUD). Both safety and efficacy of the treatment will be assessed, in particular in respect to the clinical status of the patient, i.e. prevention of graft failure and chronic GvHD and of Ebstein Barr virus (EBV) viremia for MUD patients.

The conditioning proposed combines myeloablative drugs with a favorable safety profile such as treosulfan, thiotepa (Tepadina®) and fludarabine with the intent to reduce the traditional immediate and late toxicity of busulfan and cyclophosphamide.

DETAILED DESCRIPTION:
For patients transplanted from a MRD

The primary end-point is the cumulative incidence of a combined end-point defined as the time from randomization to:

* primary and secondary graft failure,
* aGVHD II-IV,
* cGVHD,
* death, whichever occurs first.

For patients transplanted from a MUD

The primary end-point is the cumulative incidence of a combined end-point defined as the time from randomization to:

* aGVHD II-IV,
* EBV viremia, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* non malignant haematological and inherited metabolic disorders benefiting from an allogeneic HSCT conditioned with a myeloablative regimen
* Availability of a matched related donor (MRD) or Matched Unrelated Donor (MUD)
* Lansky or Karnofsky Index ≥ 60
* Inherited metabolic disorders: DQ ≥ 70 (+ MRI Loes score ≤ 9 for adrenoleukodystrophy)
* Adequate cardiac, renal, hepatic and pulmonary functions as evidenced by:
* Serum creatinine ≤ 1.5 × upper limit of normal (ULN)
* Heart shortening fraction (left-ventricle) > 28 % or LVEF > 55%
* Serum bilirubin ≤ 1.5 × ULN (except for Wolman disease),
* AST and ALT ≤ 2.5 × ULN (except for thalassemic syndromes and Wolman disease)
* Pulmonary function: if cooperative: FEV1 and FVC on pulmonary function testing > 60 %; if non cooperative: pulse oximetry > 95 % in room air
* Availability of autologous back up marrow (> 2 x 108 TNC+ cells/kg or > 2 x 106 CD34+ cells/kg) for MUD
* Adequate contraception in female patients of child-bearing potential
* Signed informed consent

Exclusion Criteria:

* Any malignancy
* Liver cirrhosis evidenced on liver histology (performed in suspicious cases or in case of Wolman disease)
* HIV- positivity
* Clinically significant pleural effusion or ascites
* Pregnancy or lactation
* Known hypersensitivity to trial drugs
* Participation in another experimental drug trial in the 2 months preceding enrollment
* Non-cooperative behaviour or non-compliance
* Previous HSCT

Ages: 28 Days to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Acute graft-versus-host disease (aGVHD) II-IV and chronic GvHD | From date of randomization assessed up to 100 months
  For patients transplanted from a MRD
  The cumulative incidence of a combined end-point defined as the time from randomization to:
  * primary and secondary graft failure,
  * aGVHD II-IV,
  * cGVHD,
  * death, whichever occurs first.
  For patients transplanted from a MUD
  The cumulative incidence of a combined end-point defined as the time from randomization to:
  * aGVHD II-IV,
  * EBV viremia, whichever occurs first.

SECONDARY OUTCOMES:
Chronic graft-versus-host disease (cGVHD) | From date of randomization assessed up to 100 months
  The cumulative incidence and severity of cGVHD
Treatment related mortality (TRM) | From date of randomization assessed up to 100 months
  The incidence of TRM
Overall survival (OS) | From date of randomization assessed up to 100 months
  The overall survival probability

CONTACTS AND LOCATIONS:
Overall Officials: Franco Locatelli, Prof, Principal Investigator — Bambino Gesù Hospital and Research Institute
Locations (4):
- Italy (4):
  - University of Cagliari, Cagliari, Italy
  - San Raffaele Scientific Institute, Milan, Italy
  - University of Milano-Bicocca San Gerardo Hospital, Monza, Italy
  - Bambino Gesù Hospital and Research Institute, Rome, Italy

REFERENCES:
- [Background] Bacigalupo A, Lamparelli T, Barisione G, Bruzzi P, Guidi S, Alessandrino PE, di Bartolomeo P, Oneto R, Bruno B, Sacchi N, van Lint MT, Bosi A; Gruppo Italiano Trapianti Midollo Osseo (GITMO). Thymoglobulin prevents chronic graft-versus-host disease, chronic lung dysfunction, and late transplant-related mortality: long-term follow-up of a randomized trial in patients undergoing unrelated donor transplantation. Biol Blood Marrow Transplant. 2006 May;12(5):560-5. doi: 10.1016/j.bbmt.2005.12.034. PMID 16635791
- [Background] Bacigalupo A, Lamparelli T, Bruzzi P, Guidi S, Alessandrino PE, di Bartolomeo P, Oneto R, Bruno B, Barbanti M, Sacchi N, Van Lint MT, Bosi A. Antithymocyte globulin for graft-versus-host disease prophylaxis in transplants from unrelated donors: 2 randomized studies from Gruppo Italiano Trapianti Midollo Osseo (GITMO). Blood. 2001 Nov 15;98(10):2942-7. doi: 10.1182/blood.v98.10.2942. PMID 11698275
- [Background] Ballet JJ, Griscelli C, Coutris C, Milhaud G, Maroteaux P. Bone-marrow transplantation in osteopetrosis. Lancet. 1977 Nov 26;2(8048):1137. doi: 10.1016/s0140-6736(77)90592-x. No abstract available. PMID 73050
- [Background] Bartelink IH, Bredius RG, Belitser SV, Suttorp MM, Bierings M, Knibbe CA, Egeler M, Lankester AC, Egberts AC, Zwaveling J, Boelens JJ. Association between busulfan exposure and outcome in children receiving intravenous busulfan before hematologic stem cell transplantation. Biol Blood Marrow Transplant. 2009 Feb;15(2):231-41. doi: 10.1016/j.bbmt.2008.11.022. PMID 19167683
- [Background] Bartelink IH, Bredius RG, Ververs TT, Raphael MF, van Kesteren C, Bierings M, Rademaker CM, den Hartigh J, Uiterwaal CS, Zwaveling J, Boelens JJ. Once-daily intravenous busulfan with therapeutic drug monitoring compared to conventional oral busulfan improves survival and engraftment in children undergoing allogeneic stem cell transplantation. Biol Blood Marrow Transplant. 2008 Jan;14(1):88-98. doi: 10.1016/j.bbmt.2007.09.015. PMID 18158965
- [Background] Basara N, Baurmann H, Kolbe K, Yaman A, Labopin M, Burchardt A, Huber C, Fauser AA, Schwerdtfeger R. Antithymocyte globulin for the prevention of graft-versus-host disease after unrelated hematopoietic stem cell transplantation for acute myeloid leukemia: results from the multicenter German cooperative study group. Bone Marrow Transplant. 2005 May;35(10):1011-8. doi: 10.1038/sj.bmt.1704957. PMID 15821768
- [Background] Bernardo ME, Zecca M, Piras E, Vacca A, Giorgiani G, Cugno C, Caocci G, Comoli P, Mastronuzzi A, Merli P, La Nasa G, Locatelli F. Treosulfan-based conditioning regimen for allogeneic haematopoietic stem cell transplantation in patients with thalassaemia major. Br J Haematol. 2008 Nov;143(4):548-51. doi: 10.1111/j.1365-2141.2008.07385.x. PMID 18986389
- [Background] Bernaudin F, Socie G, Kuentz M, Chevret S, Duval M, Bertrand Y, Vannier JP, Yakouben K, Thuret I, Bordigoni P, Fischer A, Lutz P, Stephan JL, Dhedin N, Plouvier E, Margueritte G, Bories D, Verlhac S, Esperou H, Coic L, Vernant JP, Gluckman E; SFGM-TC. Long-term results of related myeloablative stem-cell transplantation to cure sickle cell disease. Blood. 2007 Oct 1;110(7):2749-56. doi: 10.1182/blood-2007-03-079665. Epub 2007 Jul 2. PMID 17606762
- [Background] Chiesa R, Cappelli B, Crocchiolo R, Frugnoli I, Biral E, Noe A, Evangelio C, Fossati M, Roccia T, Biffi A, Finizio V, Aiuti A, Broglia M, Bartoli A, Ciceri F, Roncarolo MG, Marktel S. Unpredictability of intravenous busulfan pharmacokinetics in children undergoing hematopoietic stem cell transplantation for advanced beta thalassemia: limited toxicity with a dose-adjustment policy. Biol Blood Marrow Transplant. 2010 May;16(5):622-8. doi: 10.1016/j.bbmt.2009.11.024. Epub 2009 Dec 4. PMID 19963071